CLINICAL TRIAL: NCT06977672
Title: Effects of Down Dog Yoga on Pre-writing Skills in Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/24/0734
Record Dates: First submitted 2025-04-17; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome
Keywords: Down Dog yoga; JTHFT; BBT; pre-writing skills
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This study involves two groups of children: an experimental group (Group A) and a control group (Group B), to compare the effects of a yoga-based intervention with standard educational activities. Group A will follow a 10-week program, including an initial and final assessment, with an 8-week intervention in between. They will participate in down dog yoga sessions four times a week-two expert-led (40-45 minutes) and two parent-led (20-25 minutes). Group B will attend regular writing sessions, four times a week for 20 minutes, in small groups. Their writing will be assessed across four developmental stages: pre-phonemic, semi-phonemic, phonemic, and conventional. The study aims to evaluate developmental differences between the two approaches.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga exercise group (Experimental): This 10-week study includes assessments before and after an 8-week dog down yoga intervention. Sessions occur 3-4 times weekly, with expert-led (40-45 min) and parent-led (20-25 min) formats.
  Interventions: Other: Down Dog Yoga
- routine therapy group (Other): Children attended 20-minute group sessions four days a week for 10 weeks. Writing assessment comprised across four stages: pre-phonemic, semi-phonemic, phonemic, and conventional.
  Interventions: Other: Traditional

INTERVENTIONS:
Other: Down Dog Yoga — In this study, a period of 10 weeks, commencing with a preliminary assessment during the first week, followed by an 8-week intervention phase, and concluding with a final assessment in the last week of the study period. The frequency-intensity-time-type principle will be implemented as follows: sessions will occur 4 times per week, consisting of 2 sessions led by experts and 2 sessions involving parents. The intensity will be 40 to 45 minutes for expert-led sessions and 20 to 25 minutes for parent-led sessions. These sessions will take place 3 or 4 times per week over an 8-week period, focusing on a type of intervention known as dog down yoga
  Arms: Yoga exercise group
Other: Traditional — The children took part in group sessions four days a week over a span of 10 weeks, totaling 40 sessions. Each session, lasting around 20 minutes, involved small groups of four to seven children. The aim will be to evaluate the children's writing across four stages of development: pre-phonemic, semi-phonemic, phonemic, and conventional
  Arms: routine therapy group

SUMMARY:
Down syndrome is a genetic condition caused by an extra chromosome 21, affecting physical and cognitive development. This study will evaluate the effects of down dog yoga on prewriting skills in children with Down syndrome aged 4-8 years. A randomized controlled trial with 32 participants will be conducted at Bahawal Victoria Hospital over 10 months. Assessments will include JTHFT, BBT, and the Prewriting Skills Scale.

DETAILED DESCRIPTION:
Down syndrome is a genetic condition where people are born with an extra chromosome. Most people have 23 pairs of chromosomes within each cell in their body, for a total of 46. A person diagnosed with Down syndrome has an extra copy of chromosome 21, which means their cells contain 47 total chromosomes instead of 46. This changes the way their brain and body develop. Down syndrome causes physical, cognitive and behavioral symptoms. Down syndrome occurs in approximately 1 in 1,000 to 1 in 1,100 live births globally. Each year, around 3,000 to 5,000 children are born with this genetic condition characterized by an extra chromosome. Children with Down syndrome may experience challenges with fine motor skills because of low muscle tone or hypermobility in their hands, wrists, or elbows. This instability in their hands can significantly hinder their ability to perform advanced fine motor tasks such as prewriting, using zippers and buttons, or cutting. Early intervention refers to a structured approach involving therapy, exercises, and activities aimed at addressing developmental delays in children with Down syndrome or other disabilities. For addressing pre writing skills in Down syndrome Down dog yoga will be provided.

The study design will be Randomized Controlled Trial and will be conducted in Bahawal Victoria Hospital with the sample size of 34, age ranging 4 to 8 years. This study will be completed in time duration of 10 months after the approval of synopsis. Non-probability convenient sampling technique will be used and participants will be recruited in study after randomization. The subjects will be divided into two groups i.e one being experimental group and the other control group. Inclusion criteria will be including both genders of age group 4 to 8 years of children with down syndrome and exclusion criteria will be any deformity, injury any previous 6 month surgery. Tools will be Jebsen-Taylor Hand Function Test (JTHFT) , box and block test (BBT) and pre writing skills scale.

Reliability of JTHFT is 0.9, BBT is >0.95 and pre writing skills is 0.91 with high variability in writing performance.

ELIGIBILITY:
Inclusion Criteria:

* Children with age group 4-8years
* Both Genders (male female)
* Children who can do Independent standing and walking

Exclusion Criteria:

* Any deformity
* Pain and/or symptomatic neurologic/orthopedic dysfunction of upper or lower extremities
* Cervical injury and chest wall disorders
* Injury
* Fractures
* History of previous surgery
* Children with impaired Fun

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Jebsen-Taylor hand function test: | preliminary assessment 1 week, intervention 8 week, final assessment 1 week
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized assessment used to evaluate hand function through tasks that simulate everyday activities such as writing, feeding, and object manipulation. Commonly used in rehabilitation for individuals with neurological or musculoskeletal conditions like stroke, spinal cord injury, or hand trauma, the test consists of timed subtests that measure the speed and efficiency of hand use. It provides objective data to monitor functional ability, compare hand performance, and track rehabilitation progress.

SECONDARY OUTCOMES:
Box and block test | preliminary assessment 1 week, intervention 8 week, final assessment 1 week
  The Box and Block Test (BBT) is a quick, standardized test that measures gross manual dexterity. It involves moving as many blocks as possible from one side of a box to the other in 60 seconds, one hand at a time. It's commonly used in rehab to assess hand function in individuals with neurological conditions.
  The Box and Block Test (BBT) is a quick, standardized test that measures gross manual dexterity. It involves moving as many blocks as possible from one side of a box to the other in 60 seconds, one hand at a time. It's commonly used in rehab to assess hand function in individuals with neurological conditions.

OTHER OUTCOMES:
Pre writing skills | preliminary assessment 1 week, intervention 8 week, final assessment 1 week
  Pre-writing skills are the foundational motor and cognitive abilities children develop before learning to write. These include fine motor control, pencil grip, hand-eye coordination, and the ability to draw basic shapes. They are essential for building the strength and coordination needed for writing letters and numbers effectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yusra Uzlifat, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields N. Physiotherapy management of Down syndrome. J Physiother. 2021 Oct;67(4):243-251. doi: 10.1016/j.jphys.2021.08.016. Epub 2021 Sep 10. No abstract available. PMID 34511385